CLINICAL TRIAL: NCT00233350
Title: Clinical Evaluation of Navigated 3D Ultrasound Multicentre Study
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Multicentre_3DUS
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2012-10

CONDITIONS: Brain Neoplasms
Keywords: Neuronavigation; Ultrasound; Brain tumour surgery; Biopsy; Histopathology; Intraoperative imaging; 3D ultrasound imaging
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: use of navigated 3D ultrasound during surgery

SUMMARY:
3D ultrasound is a new modality used in image guided neurosurgery. a multicentre study is started for the evaluation of this tool as a means for achieving total resection of brain tumors at greater safety.

DETAILED DESCRIPTION:
The degree of resection as judged by the surgeon is recorded at the end of surgery for each patient, and then compared with the postoperative MRI. Neurological status before and after surgery, QOL before surgery and at follow-up as well as survival is recorded.

ELIGIBILITY:
Inclusion Criteria:

* Supratentorial glioma

Exclusion Criteria:

* Not willing to participate in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were operated for intracranial high-grade gliomas (World Health Organisation(WHO) grade III/IV) in the 3-year period between January 1st 2007 and December 31st 2009 in the Department of Neurosurgery, St. Olavs University Hospital, Trondheim, Norway
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geirmund Unsgaard, MD, PhD, Study Director — National Taiwan Normal University
Locations (1):
- St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Solheim O, Selbekk T, Jakola AS, Unsgard G. Ultrasound-guided operations in unselected high-grade gliomas--overall results, impact of image quality and patient selection. Acta Neurochir (Wien). 2010 Nov;152(11):1873-86. doi: 10.1007/s00701-010-0731-5. Epub 2010 Jul 21. PMID 20652608